CLINICAL TRIAL: NCT00720668
Title: The Risk of Exacerbation of Chronic Hepatitis B After Percutaneous Radiofrequency Ablation of Hepatocellular Carcinoma
Acronym: HBV-HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: minshan chen, cancer canter, Sun Yat-sen University
Other Study IDs: RFA006
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Hepatitis B; Hepatocellular Carcinoma
Keywords: hepatitis B; hepatocellular carcinoma; radiofrequency ablation; reactivation
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patient with hepatocellular carcinoma after radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — radiofrequency ablation for HCC
  Other Names: RFA

SUMMARY:
This study aim to find out the risk of exacerbation of chronic hepatitis B after percutaneous radiofrequency ablation (RFA) or hepatectomy for HCC, and it's effect to treatment outcome.

DETAILED DESCRIPTION:
It has been reported that HBV replication can be reacted after chemotherapy or immunotherapy, which will lead to exacerbation of chronic hepatitis B (ECHB). It is still unknown that if percutaneous radiofrequency ablation or liver resection for hepatocellular carcinoma (HCC) will react the replication of HBV or not. This study aim to find out the risk of exacerbation of chronic hepatitis B after percutaneous radiofrequency ablation (RFA) or hepatectomy for HCC, and it's effect to treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* HBV carrier with HCC
* After percutaneous radiofrequency ablation;
* No history of encephalopathy, ascites refractory to diuretics or variceal bleeding
* No HCV or HIV co-infection
* No previous treatment of HCC
* No previous treatment of HBV except Lamivudine

Exclusion Criteria:

* Patient compliance is poor
* Active clinically serious infections ( > grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Distantly extrahepatic metastasis
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Excluded therapies and medications, previous and concomitant
* Prior use of any systemic anti-cancer treatment for HCC, eg. chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior randomization
* Prior use of systemic investigational agents for HCC
* Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatocellular carcinoma (HCC) after percutaneous radiofrequency ablation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-03 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The Rate of Exacerbation of chronic hepatitis B after RFA | one week, one month, one year

SECONDARY OUTCOMES:
survival | 1, 3, 5-year
mortality | one month

CONTACTS AND LOCATIONS:
Overall Officials: min-shan chen, MD, Principal Investigator — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Result] Poon RT, Fan ST, Tsang FH, Wong J. Locoregional therapies for hepatocellular carcinoma: a critical review from the surgeon's perspective. Ann Surg. 2002 Apr;235(4):466-86. doi: 10.1097/00000658-200204000-00004. PMID 11923602
- [Result] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695